CLINICAL TRIAL: NCT05154305
Title: Multidisciplinary Rehabilitation of Children and Adolescents After Acute Cancer Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: VZW kinderkankerfonds, Belgium (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018/0709
Record Dates: First submitted 2021-11-29; First posted 2021-12-13 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Cancer Survivors; Rehabilitation; Exercise Therapy
Keywords: Multidisciplinary Rehabilitation; Cohort study; Childhood and adolescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children 6 months post acute treatment (Experimental): children and adolescents between 6 months and 8 years post acute cancer treatment
  Interventions: Behavioral: multidisciplinary intervention

INTERVENTIONS:
Behavioral: multidisciplinary intervention — * individually adjusted physical program consisting of strength and endurance training > 3 times a week, 2 times guided by a physical therapist at the University Hospital or at a private practice, and ones a week by themselves at home recorded by an activity tracker. Follow-up is foreseen on monthly basis.
  * multidisciplinary coaching (discipline depending on personal needs of patient) on a monthly basis. These coaching sessions could be in small groups or individual.

SUMMARY:
Recent numbers display a 85% survival-rate in children after a very harmful disease such as cancer. However, the survivors still experience mild to severe side effects of the primary disease or treatment.

A long time follow-up in the University Hospital of Ghent in children with cancer displays important long term side effects such as: reduced muscle strength; reduced endurance capacity; reduced exercise tolerance; fatigue; disturbed body composition with increased risk for obesity and/or diabetes and osteoporosis; and neuropathic damage and myopathy. These physical complaints have a significant impact on the activities and participation in daily living.

The purpose of this interventional study is to create a rehabilitation program for children after acute cancer treatment. The goal is to minimalize the previous described long term side effects of the disease. The current study should allow us to determine the effects of the intervention at the level of functioning, activities and participation. In addition, we account for the environment and personal factors as described by the International Classification of Functioning, disability and health (ICF-criteria).

The study population consists of children between 8 and 11 years and adolescents of 12 to 21 years old. All participants receive a multidisciplinary treatment for 4 months, guided by a team which includes: oncologist, rehabilitation doctor, physical therapist, dietitian, psychologist, and occupational therapist.

At the beginning of the multidisciplinary program, the participants receive psychoeducation, diet advice, tips for participation, fatigue, and psychological well-being. In general, the rehabilitation program focusses on reintegration at school and leisure activity.

After the first assessment, an individually adjusted physical program consisting of strength and endurance training will be made. This physical program will be executed 3 times a week, 2 times guided by a physical therapist at the University Hospital or at a private practice, and ones a week by themselves at home recorded by an activity tracker. Follow-up is foreseen on monthly basis.

Participants will undergo assessment 3 times: 1) baseline (T0); 2) after 4 months treatment (T1); 3) after 1 year follow-up (T2).

The purpose of this program is to encourage patients at risk for increasing their healthy habits, exercise and participation in order to decrease long-term (side) effects.

ELIGIBILITY:
Inclusion Criteria:

* between 6 months and 8 years post acute cancer treatment
* off medical treatment
* all possible cancer diagnosis, except for brain tumors and sarcomas

Exclusion Criteria:

* not able to participate for 3 consecutive weeks
* not able to perform a maximal cardiopulmonary exercise test
* unwilling to cooperate
* relapse

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximal exercise test | 20 minutes
  Maximal exercise test on a cycle ergometer
Body composition | 5 minutes
  Body composition by dietitian
Pediatric Quality of Life Inventory | 10 minutes
  assessment Quality of Life
Children's Assessment of Participation and Enjoyment (CAPE) | 10 minutes
  assessment participation
Preferences for Activities of Children (PAC) | 10 minutes
  assessment preferred activities

CONTACTS AND LOCATIONS:
Overall Officials: Catharina Dhooghe, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chamorro-Vina C, Ruiz JR, Santana-Sosa E, Gonzalez Vicent M, Madero L, Perez M, Fleck SJ, Perez A, Ramirez M, Lucia A. Exercise during hematopoietic stem cell transplant hospitalization in children. Med Sci Sports Exerc. 2010 Jun;42(6):1045-53. doi: 10.1249/MSS.0b013e3181c4dac1. PMID 19997035
- [Background] Huang TT, Ness KK. Exercise interventions in children with cancer: a review. Int J Pediatr. 2011;2011:461512. doi: 10.1155/2011/461512. Epub 2011 Oct 27. PMID 22121378
- [Background] Kelly AK. Physical activity prescription for childhood cancer survivors. Curr Sports Med Rep. 2011 Nov-Dec;10(6):352-9. doi: 10.1249/JSR.0b013e318237be40. PMID 22071396
- [Background] Kotte EM, DE Groot JF, Bongers BC, Winkler AM, Takken T. Validity and Reproducibility of a New Treadmill Protocol: The Fitkids Treadmill Test. Med Sci Sports Exerc. 2015 Oct;47(10):2241-7. doi: 10.1249/MSS.0000000000000657. PMID 26378949
- [Background] San Juan AF, Wolin K, Lucia A. Physical activity and pediatric cancer survivorship. Recent Results Cancer Res. 2011;186:319-47. doi: 10.1007/978-3-642-04231-7_14. PMID 21113771
- [Background] Stark T, Walker B, Phillips JK, Fejer R, Beck R. Hand-held dynamometry correlation with the gold standard isokinetic dynamometry: a systematic review. PM R. 2011 May;3(5):472-9. doi: 10.1016/j.pmrj.2010.10.025. PMID 21570036
- [Background] Steinberg A, Asher A, Bailey C, Fu JB. The role of physical rehabilitation in stem cell transplantation patients. Support Care Cancer. 2015 Aug;23(8):2447-60. doi: 10.1007/s00520-015-2744-3. Epub 2015 May 14. PMID 25971213
- [Background] van Dijk-Lokkart EM, Braam KI, Huisman J, Kaspers GJ, Takken T, Veening MA, Bierings M, Merks JH, Grootenhuis MA, van den Heuvel-Eibrink M, Streng IC, van Dulmen-den Broeder E. Factors influencing childhood cancer patients to participate in a combined physical and psychosocial intervention program: Quality of Life in Motion. Psychooncology. 2015 Apr;24(4):465-71. doi: 10.1002/pon.3677. Epub 2014 Oct 6. PMID 25285989
- [Background] West SL, Gassas A, Schechter T, Egeler RM, Nathan PC, Wells GD. Exercise intolerance and the impact of physical activity in children treated with hematopoietic stem cell transplantation. Pediatr Exerc Sci. 2014 Aug;26(3):358-64. doi: 10.1123/pes.2013-0156. Epub 2014 Apr 10. PMID 24721685
- [Background] Winter C, Muller C, Brandes M, Brinkmann A, Hoffmann C, Hardes J, Gosheger G, Boos J, Rosenbaum D. Level of activity in children undergoing cancer treatment. Pediatr Blood Cancer. 2009 Sep;53(3):438-43. doi: 10.1002/pbc.22055. PMID 19415742
- [Background] BONGERS, B.C., VAN BRUSSEL, M., HULZEBOS, E.H.J. & TAKKEN, T. (2014). PEDIATRIC NORMS FOR CARDIOPULMONARY EXERCISE TRAINING: IN RELATION TO SEX AND AGE (2ND ED.). UTRECHT: BOXPRESS.
- [Background] TAKKEN, T., VAN BRUSSEL, M., HULZEBOS., H.J., (2008). INSPANNINGSFYSIOLOGIE BIJ KINDEREN. HOUTEN: BOHN STAFLEU VAN LOGHUM.
- See also: project description on sponsor's website — https://www.kinderkankerfonds.be/projecten-en-activiteiten/kaboost/